CLINICAL TRIAL: NCT05440916
Title: Palliative RadIotherapy of Multiple Metastatic Sites Before First Line of Systemic Therapy With Immune Checkpoint Inhibitors and Chemotherapy in Metastatic Non-Small-Cell Lung Cancer (PRIMM Study)
Brief Title: Palliative RadIotherapy of Multiple Metastatic Sites Before First Line of Systemic Therapy With Immune Checkpoint Inhibitors and Chemotherapy in Metastatic Non-Small-Cell Lung Cancer
Acronym: PRIMM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Collaborators: Institute of Oncology Ljubljana (Other); The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Tanja Znidaric Rakar, Principal Investigator, University Medical Centre Maribor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0120-127/2022/3
Record Dates: First submitted 2022-05-30; First posted 2022-07-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Metastatic Lung Non-Small Cell Carcinoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients with metastatic Non-Small Cell Lung Carcinoma eligible for first line systemic treatment with chemotherapy and immune checkpoint inhibitors (PDL1 less than 50%)
  Radiotherapy: palliative irradiation of 2 to 5 sites (parenchymal/bone/soft tissue metastasis and/or primary lung tumour) with fractionation: 5 fractions of 4Gy (total dose 20Gy) in one week before systemic therapy.
  Interventions: Radiation: Palliative Radiotherapy: 5 x 4Gy; Drug: chemotherapy + immune checkpoint inhibitors
- Historical cohort (Other): Patients with metastatic Non-Small Cell Lung Carcinoma treated with first line of systemic therapy with chemotherapy and immune checkpoint inhibitors (PDL1 less than 50%).
  Radiotherapy: no radiation therapy during the first line of systemic treatment before progression of disease.
  Interventions: Drug: chemotherapy + immune checkpoint inhibitors

INTERVENTIONS:
Radiation: Palliative Radiotherapy: 5 x 4Gy — Palliative irradiation of 2 to 5 sites (metastatic sites or/and primary lung tumour) in one week before systemic therapy. Systemic therapy should be given as soon as possible after irradiation.
  Arms: Study group
Drug: chemotherapy + immune checkpoint inhibitors — Systemic therapy according to national/European recommendations.

SUMMARY:
The study is designed as a non-randomized Phase 2 clinical intervention study. The study will include patients with disseminated Non-Small Cell Lung Carcinoma (NSCLC) which are eligible for first line of systemic treatment with immune checkpoint inhibitors and platinum-based chemotherapy (PDL1 less than 50%). Patients will receive palliative radiotherapy to multiple sites (2 to 5 sites) prior to systemic treatment.

Results of treatment will be compared to historical cohort of patients treated only with systemic therapy.

DETAILED DESCRIPTION:
The primary objective is to investigate efficacy of radiation therapy before the first line of systemic therapy with immune checkpoint inhibitors and platinum-based chemotherapy in metastatic NSCLC (PDL1 less than 50%).

ELIGIBILITY:
Inclusion Criteria:

* Signed consent to the study before the start of the procedures related to the protocol
* Age ≥ 18 years at time of study entry
* ECOG performance status 0-2
* Histologically or cytologically confirmed non-small cell lung cancer, with expression of PD-L1 of less than 50%
* Stage IV metastatic Non-Small Cell Cancer confirmed by CT scan (of brain, chest and abdomen) or PET CT
* Patients must be eligible for first line of systemic treatment with standard of care checkpoint inhibitor immune therapy and chemotherapy - according to the recommendations
* inclusion of patients treated for few brain metastases (with surgery or ablative radiosurgery) is permitted (if the disease in the central nervous system is under control)
* Prior surgery (diagnostic and therapeutic) and irradiation (for example: stereotactic irradiation of brain metastases) is permitted, provided that patients have fully recovered from the procedure at least 2 weeks before inclusion in the study
* Patients treated with surgery or radiation and chemotherapy for limited non-small cell carcinoma in the past is permitted

Exclusion Criteria:

* Metastatic non-small cell carcinoma with known oncogenic alterations suitable for targeted treatment
* Brain or meningeal metastases that are not under control
* Other malignancy (other than non-small cell carcinoma) present that has progressed and/or requires active treatment
* Previous malignancy, unless cured or complete remission has been achieved for at least 2 years prior to enrolment and does not require maintenance treatment. With the exception of basal cell carcinoma or squamous cell carcinoma of skin, which was treated and precancerous diseases and in situ cancers
* Patients with interstitial lung disease
* The possibility of radical treatment of oligometastatic disease (primary tumour and metastases)
* Patients who are not eligible for checkpoint immune inhibitor treatment due to contraindications such as autoimmune diseases, with the exception of some exceptions (Vitiligo; type I diabetes; hormone replacement hypothyroidism; psoriasis that does not require systemic treatment or other autoimmune diseases that do not limit checkpoint immune inhibitors treatment)
* Previous treatment with anti PD-1, anti PD-L1, anti CTLA-4 antibodies, or any other treatment that affects T lymphocytes or checkpoint pathways
* Patients with known sensitivity to monoclonal antibodies
* Patients with known HIV infection
* Patients with active or chronic hepatitis B and / or C
* Pregnant and breastfeeding mothers
* Patients with serious and uncontrollable health problems (physical and mental), which, according to researchers, could affect the poor participation of patients and make it difficult to interpret the results
* Patients on corticosteroid therapy (more than 10 mg methylprednisolone or equivalent) prior to enrolment
* Irradiation 2 months before inclusion in the study, except for stereotactic irradiation of brain metastases (or radiation and chemotherapy for limited non-small cell carcinoma in the past)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months after the completion of study.
  Disease status will be evaluated based on imaging results until progression or death; assessed every three months.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of randomization until the date of death, or the last follow up date on which the participant was reported alive, assessed up to 18 months.
  Amount of time from treatment until death, reported via follow up visit or phone call.
Objective Response Rate (ORR) | Assessment after 3 months after the date of randomization and every 3 months up until progression. Assessed up to 18 months after the completion of study.
  Using assessment according to RECIST (after 3 months and time to ORR). Percentage of patients with a complete response or partial response.
Patterns of progression | Assessed up to 18 months after the completion of study.
  Percentage of patients with recorded first site of progression of disease at irradiated sites and non-irradiated sites or both.
A review of predictive maker PDL1 - indicating a better response to combination therapy | From the start of treatment until the date of documented progression or death, whichever comes first, assessed up to 18 months after the completion of study.
  - Percentage of PDL 1 expression on tumour cells, where PFS was significantly better in combination therapy.

CONTACTS AND LOCATIONS:
Locations (3):
- Slovenia (3):
  - University Clinic Golnik, Golnik
  - Institute of Oncology Ljubljana, Ljubljana
  - University Medical Centre Maribor, Maribor

IPD SHARING:
Plan to Share IPD: No